CLINICAL TRIAL: NCT04245761
Title: Pilot Open Non-Comparative Study To Evaluate In Special Care Setting The Administration Of A New Nutraceutical Associated With Sleep Hygiene Guidelines In Subjects Affected By Persistent Mild Sleep Disorders
Brief Title: Open Non-Comparative Study To Evaluate Administration Of a New Nutraceutical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Italfarmaco (Industry)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS/18/SON/01
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Pilot, open, non-comparative, multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonidor® (Experimental): Application: following the summary of product characteristics (l tablet per day) At the 7-day phone call the Investigator can increase the dosage to 2 tablets per day only in non-responding subjects.
  Interventions: Dietary Supplement: Sonidor®

INTERVENTIONS:
Dietary Supplement: Sonidor® — Sonidor® triple layer release tablets are developed with a specialized process to improve stability and bioavailability of the formulation based on hawthorn, lavender and hop extracts. The hawthorn, lavender and hop extracts used to product Sonidor® have an elevated content of vitexin (3%), monoterpens (4% as linalool) and flavonoids (4%), respectively.

SUMMARY:
The Research Hypothesis for the present pilot study in a special care setting is that in a population suffering of mild and recent sleep disorders the pre-sleep arousal measured by the Pre-Sleep Arousal Scale (PSAS) after 30 days of oral administration with a nutraceutical composed of hawthorn, lavender and hop (Sonidor®) shall significantly improve in comparison with the baseline condition.

DETAILED DESCRIPTION:
Sonidor® was developed as a nutraceutical composed of hawthorn, lavender and hop inducing sleep and relaxation in subjects with mild sleep disturbances. In addition, the Sonidor® innovative three-layer-tablet formulation should allow the active components to be released with different speeds into the gastrointestinal tract exerting a synergistic action to induce sleep-promoting effects.

Primary objective is to have a preliminary evaluation of the efficacy of Sonidor® in subjects affected by persistent mild sleep disorders (difficulty in initiating sleep for at least 1 month and reduced quality of sleeping) to whom in special care setting have been suggested sleep hygiene guidelines and administered the tested nutraceutical for one month.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 to 70 years with persistent, recent (at least 1 month) and mild sleep disorders related to pre-sleep arousal and reduced quality of sleeping;
2. PSAS at baseline between 16 and 24;
3. ISI at baseline ≥ 12;
4. Able to communicate adequately with the Investigator and to comply with the requirements for the entire study;
5. Capable of and freely willing to provide written informed consent prior to participating in the study;

Exclusion Criteria:

l. Subjects with Morningness-Eveningness Questionnaire Self-Assessment (MEQSA) values between 16 and 41; 2. Pregnancy and/or breast-feeding; 3. Subjects assuming beta blockers, hypnotic or sedative drugs or other nutraceuticals; 4. Psychosis, schizophrenia, mania, depressive disorders, history of suicide attempt, or suicidal ideation, or any other psychiatric illness (with the exception of intermittent anxiety); 5. Known intolerance to the tested product or at one of the ingredients (hawthorn, lavender or hop); 6. Drug or alcohol abuse within 12 months of Day 0; 7. All clinical conditions that, at the evaluation of the Investigator, can be referred to as secondary insomnia; 8. Participation in an interventional clinical study or administration of any investigational agents in the previous 30 days; 9. Presence of any clinically significant medical condition judged by the investigator to preclude the subject's inclusion in the study;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Pre-sleep arousal scale (PSAS); | 30 days
  Change in Pre-sleep arousal scale PSAS from a maxim of 24 to a minimum of 16 is a positive outcome for the investigational product

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | 30 days
  Minimal score for ISI scale is 0 to 7 (clinical insignificant insomnia), 8 to 14 (bellow average insomnia), 15 to 21 (moderate insomnia) and 22 to 28 (severe insomnia)
Patient Health Questionnaire QoL (PHQ-9) | 30 days
  The minimal score of this questionnaire is 0 (patient is not affected by insomnia) and the maximum score is 27 ( patient is highly affected by insomnia)
Cognitive subscale of Pre-sleep arousal scale (PSAS) | 30 days
  The minimal score of this questionnaire is 0 (patient is not affected by insomnia) and the maximum score is 27 ( patient is highly affected by insomnia)
Somatic subscale of PSAS (Pre-sleep arousal scale) | 30 days
  The minimal score of this questionnaire is 0 (patient is not affected by insomnia) and the maximum score is 27 ( patient is highly affected by insomnia)
Global Assessment of Safety | 30 days
  it will be reported by the subject using the 4-point scale: 1= very good safety, 2 = good safety, 3 = moderate safety and 4 = poor safety. Global Assessment of Safety will be evaluated at the last visit.
Restorative Sleep Questionnaire-Daily (RSQ-D) | 30 days
  Provides a valid and reliable measure for assessing nonrestorative sleep complaints. It includes 9 self-report items related to various aspects of the restorative quality of sleep. The paper printed questionnaire will be completed on a daily basis by subject upon awakening. Minimum score is 0 and maximum is 100. The higher the score, the better the sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Turcu, Principal Investigator — Fizio Center
Locations (1):
- Fizio Center, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No